CLINICAL TRIAL: NCT05572801
Title: NOAC9 - A Phase II Randomised Nordic Anal Cancer Group Study on Circulating Tumor DNA Guided Follow-Up
Brief Title: NOAC9 - Circulating Tumor DNA Guided Follow-Up in Anal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Comprehensive Cancer Center (Other); Nordic Cancer Union (Other); The regions medicine- and treatment funds (Unknown)
Responsible Party: Principal Investigator, Karen-Lise Garm Spindler, Professor, Dr. Med., Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 82386
Record Dates: First submitted 2022-08-22; First posted 2022-10-10 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anal Cancer
Keywords: Anal cancer; Circulating Tumor DNA; Plasma HPV; Follow-up
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A: HPV positive standard of care follow-up (No Intervention): The national follow-up program + collection of blood samples for retrospective translational research
- ARM B: HPV positive ctDNA guided imaging in follow-up (Experimental): The national follow-up program + ctDNA guided additional imaging + collection of blood samples for retrospective translational research
  Interventions: Diagnostic Test: AMR B: HPV positive ctDNA guided imaging in follow-up
- ARM O: HPV negative observational arm (No Intervention): Patients with HPV negative disease will be included in an observational arm (ARM O)
  ARM O: The national follow-up program + collection of blood samples for retrospective translational research

INTERVENTIONS:
Diagnostic Test: AMR B: HPV positive ctDNA guided imaging in follow-up — Blood samples in follow-up positive for ctDNA leads to an extra PET-CT scan to detect early treatment failure
  Arms: ARM B: HPV positive ctDNA guided imaging in follow-up

SUMMARY:
This study investigates if circulating tumor DNA can improve the detection of early treatment failure or recurrence in localized squamous cell carcinoma of the anus (SCCA) after curative chemoradiotherapy thereby increasing the potential for cure. This will be done by comparing the standard follow-up program with ctDNA guided imaging follow-up. Secondly, the aim is to establish early interventions against late morbidities.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the anus (SCCA) is a rare disease with less than 200 new cases in Denmark and Sweden each year and approximately 100 new cases in Norway and Finland but with increasing incidence. Primary treatment is chemo-radiotherapy (CRT) comprising high dose IMRT based radiation therapy with combination chemotherapy of 5-FU and Cisplatin. Overall treatment response is good in small tumors, but less pronounced for high-risk tumors.

In absence of complete pathological response after CRT or local recurrence, patients are evaluated for. salvage surgery. The importance of R0 resection on overall survival has been described in several studies. It is suggested that early detection of treatment failure and recurrences increases the chance of possible curative surgery (R0-resection) and thereby overall survival.

A follow-up program has 3 purposes

1. To detect lack of complete response to primary treatment
2. Early detection of local or distant recurrences
3. Describing and managing late morbidity

Purpose:

The main purpose of this follow-up study is to investigate if circulating tumor tDNA can improve detection of early treatment failure or recurrences thereby assisting in increasing the potential for cure. Secondly, to provide evidence for use of imaging and third objective is to establish early intervention against late morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCCA eligible for definitive (chemo)radiotherapy
* ≥ 18 of years
* Written and oral consent

Exclusion Criteria:

* Conditions that will contraindicate blood samples
* Conditions that will contraindicate a PET-CT scan.
* Potential lack of compliance to standard FU program and study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | after 2 years
  Disease free survival 2 years from end of therapy

SECONDARY OUTCOMES:
Time between ctDNA detected and CT verified recurrences | after 5 years
  Lead time between ctDNA detected and CT verified recurrences
Rate of succesful salvage surgery | after 5 years
  Rate of succesful salvage surgery
Pattern of failure | after 5 years
  Pattern of failure defined as ln-field failures (within GTV-T, GTV-N, CTV or irradiated areas) or out-of-field failures
Disease free survival at 5 years follow-up | after 5 years
  Disease free survival at 5 years follow-up
The rate of distant failures | after 5 years
  The rate of distant failures
Overall survival | 5 years
  Overall survival from beginning of treatment to death of any cause
Explorative analysis of total circulating free DNA (cfDNA) | 5 years
  Explorative analysis of total circulating free DNA (cfDNA)
ctDNA assays for HPV negative cases | 5 years
  Analysis of ctDNA in HPV negative cases
Acute toxicity | after 2 and 5 years
  Acute toxicity (CTCAE 5.0)
Late toxicity | after 2 and 5 years
  Late toxicity (CTCAE 5.0)
Health related quality of life | after 2 and 5 years
  Health related quality of life (EORTC QLQ-ANL27)

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, Professor, Principal Investigator — Department of Experimental Clinical Oncology Aarhus Univeristy Hospital
Locations (13):
- Denmark (3):
  - Department of Oncology Herlev and Gentofte Hospital, Herlev, Capital Region of Denmark
  - Department of Oncology, Vejle Hospital, Vejle, The Regions of Southern Denmark
  - Aarhus University Hospital, Aarhus
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olav's University Hospital, Trondheim
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital Lund, Lund
  - Karonlinska University Hospital, Stockholm
  - Norrlands University Hospital, Umeå